CLINICAL TRIAL: NCT03045302
Title: A Phase IIa, Open-label, Single-arm, Two Stage, Multi-centre Study to Investigate the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of Repeated Subcutaneous Administration of BIM23B065 in Subjects With Acromegaly
Brief Title: Assessment of BIM23B065, Given as Repeated Subcutaneous Injection in Subjects With Acromegaly
Acronym: DOPAACRO 002
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination is a sponsor decision. No new safety signal or serious adverse event has been observed.
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-FR-10380-002; 2015-003868-37 (EudraCT Number)
Record Dates: First submitted 2016-11-10; First posted 2017-02-07 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — BIM23B065

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIM23B065 (Experimental)
  Interventions: Drug: BIM23B065

INTERVENTIONS:
Drug: BIM23B065 — Subcutaneous twice a day or three times a day administration of BIM23B065. Dose will be 0.4, 0.6, 0.8 or 1 mg (twice a day or three times a day).

SUMMARY:
The purpose of the protocol is evaluate the safety, the pharmacodynamics and the pharmacokinetic of repeated administration of BIM23B065 in subjects with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent prior to any study related procedures.
* Subjects will have a documented diagnosis of acromegaly.
* Subjects will have active acromegaly confirmed by a mean serum concentration of GH over 2 hours > 2.5 µg/L at screening analysed by central laboratory.
* Subjects who have had pituitary surgery must be >8 weeks post-surgery.
* 18 to 75 years of age.
* Negative pregnancy test (female subjects).
* Female who is either of non-childbearing potential or who is not pregnant at screening and agrees to use highly effective contraception during whole duration of the study. Non-childbearing potential is defined as being postmenopausal for at least 1 year, or women with documented infertility (natural or acquired).
* Male subjects must agree that, if their partner is at risk of becoming pregnant, they will use a medically accepted, effective method of contraception (i.e. condom) for the duration of the treatment period of the study.

Exclusion Criteria:

* The subject has received long-acting Somatostatin Analogues (SSA) within 12 weeks prior screening (e.g.octreotide long acting release (LAR), lanreotide Autogel, pasireotide LAR).
* The subject has received short-acting SSA within 1 week (e.g. octreotide SC) prior to screening.
* The subject has received a dopamine agonist within 6 weeks (e.g., bromocriptine or cabergoline) prior to screening.
* The subject has received GH antagonist within 12 weeks prior to screening (e.g., pegvisomant).
* The subject had undergone radiotherapy to the pituitary gland at any time prior to study entry.
* It is anticipated that the subject will undergo pituitary surgery or radiation to the pituitary gland during the study, or will require additional medical therapy for acromegaly (including SSA, pegvisomant, or dopamine agonists) during the study.
* The subject has unsubstituted/untreated adrenal insufficiency.
* If the subject has any history of postural hypotension or evidence of postural hypotension at screening (>= 20 mm Hg decrease in Systolic blood pressure (SBP), >= 10 mm Hg decrease in diastolic blood pressure, or >=30 bpm increases in pulse rate, after standing for 2 minutes from resting supine position of at least 10 min).
* Subject with poorly controlled diabetes mellitus (presence of ketoacidosis or a glycosylated hemoglobin level >10%).
* Subject with diabetes treated with insulin for less than 6 weeks prior to study entry, or with an unstable insulin dose in the 6 weeks prior to study entry or HbA1c>10%.
* Subject is taking beta-blockers (which can inhibit compensatory increases in HR during hypotensive episodes).
* Subject is being treated for hypertension and in the opinion of the investigator their antihypertensive medication puts them at increased risk of postural hypotension.
* Subject is hypotensive at screening as defined as systolic < 90 mmHg and/or diastolic <60 mmHg.
* Subject has clinically significant hepatic abnormalities and/or alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥2 x ULN and/or alkaline phosphatase (AP) ≥2 x ULN and/or total bilirubin ≥1.5 x ULN and gamma-glutamyl transferase (GGT) ≥2.5 x ULN during the Screening period (local laboratory results).
* Subject has a compression of the optic chiasm causing visual-field defects.
* Subject is receiving any oestrogen-containing Hormone Replacement Therapy (HRT).
* Subject has clinically significant pancreatic abnormalities and/or amylase and/or lipase ≥2 x ULN during the Screening period (local laboratory results).
* Any significant renal abnormalities, including confirmed proteinuria and/or creatinine ≥1.5x ULN during screening assessed by the local laboratory.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-06-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Study Director, Study Director — Ipsen
Locations (6):
- CHU de Liège, University of Liège, Domaine Universitaire du Sart-Tilman, Liège, Belgium
- Medical Centre, University of Pecs, I Department of Internal Medicine, Pécs, Hungary
- Clinical Center of Serbia, Clinic for Endocrinology, Diabetes and Metabolic Diseases, Belgrade, Serbia
- Ukraine (3):
  - "Institute of Endocrinological Pathology named after Danilevskij V.Ya., AMS of Ukraine", Department of General Endocrinology, Kharkiv
  - "Institute of Endocrinology and Metabolism named after V.P.Komisarenko, AMS Ukraine", Department of General Endocrinology, Kiev
  - Vinnitsa Regional Endocrinology Dispensary, Vinnitsa National Medical University named after M.I Pirogov, Therapeutic Department № 2, Vinnitsa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with acromegaly were recruited from 26 January 2017 in 4 study centres in 4 countries. Stage 1 of the study consisted of a twice daily (BID) regimen of BIM23B065, and a Stage 2 with a three times daily regimen of BIM23B065 was planned but not conducted due to early termination of the study on 26 May 2017.
Pre-assignment Details: 7 subjects were screened and 3 failed screening (1 subject did not meet eligibility criteria and 2 subjects did not complete screening procedures due to the early study termination).
Groups:
- BIM23B065 BID Stage 1: Subjects received twice daily administrations of BIM23B065 (at an interval of 12 +/- 1 hour) as subcutaneous injections in the abdominal region during the Stage 1 treatment period which consisted of a titration phase and a treatment phase.
  Titration phase (Days 1 to 6): Subjects received BIM23B065 0.4 milligram (mg) BID (Days 1 and 2, then BIM23B065 0.6 mg BID (Days 3 and 4) and BIM23B065 0.8 mg BID (Days 5 and 6).
  Treatment phase (Days 7 to 14): Following titration, a stable target dose of 1.0 mg BID BIM23B065 was planned to be administered from Day 7 to Day 14.
Period: Overall Study
Arm/Group | BIM23B065 BID Stage 1
Started | 4
Completed | 3
Not Completed | 1
Not completed — Pre-treatment adverse event | 1

BASELINE CHARACTERISTICS:
Population: The Intent to treat population consisted of all subjects with at least 1 BIM23B065 administration.
Arm/Group | BIM23B065 BID Stage 1
Number analyzed (Participants) | 4
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.0 (15.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: The Number of Subjects Who Were Growth Hormone (GH) Responders at Day 14 of the Treatment Period
Description: A GH responder was defined as a subject with mean serum GH concentration ≤2.5 micrograms per litre (mcg/L) or >50% reduction from mean baseline GH concentration after a 6-day titration and an 8-day treatment period with BIM23B065. The mean serum concentration of GH was measured over 6 hours at baseline (Day -1) and on Day 14. The number of subjects who were GH responders at Day 14 of the treatment period is presented.
Time Frame: From baseline (Day -1) to Day 14.
Population: The Efficacy Evaluable population consisted of all subjects with at least 1 BIM23B065 administration with available pharmacodynamic (PD) data and no protocol deviations with relevant impact on PD data, who had an evaluable primary efficacy endpoint (mean concentration of GH over 6 hours) at baseline and at Day 14.
Measure: Count of Participants; unit: Participants
Arm/Group | BIM23B065 BID Stage 1
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events were collected from Day 1 of the treatment period up to the end of Week 4 (approximately 28 days).
Description: The Safety population consisted of all subjects with at least 1 BIM23B065 administration.
Arm/Group | BIM23B065 BID Stage 1
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIM23B065 BID Stage 1 (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The sponsor stopped the study early as the preliminary results in 3 subjects dosed with BIM23B065 showed an inadequate PD profile and efficacy. The enrolled subjects only received BID treatment. Only the primary endpoint results are reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/02/NCT03045302/Prot_000.pdf
  • Statistical Analysis Plan (2017-02-10): https://cdn.clinicaltrials.gov/large-docs/02/NCT03045302/SAP_001.pdf